CLINICAL TRIAL: NCT04756765
Title: A Phase 2 Clinical Trial of Talazoparib Monotherapy for PALB2 Mutation Associated Advanced Breast Cancer
Brief Title: Talazoparib Monotherapy in PALB2 Mutation Associated Advanced Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to changes in the treatment landscape, the study faced significant recruitment challenges. As no patients were enrolled, the sponsor requested study closure
Sponsor: Stanford University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-59141; BRS0126 (Other: OnCore); NCI-2023-01961 (Registry Identifier: National Cancer Institute: Clinical Trials Reporting Program)
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Advanced Breast Cancer
Keywords: PALB2 mutation
MeSH Terms: conditions — Breast Neoplasms | interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Talazoparib Arm (Experimental): Talazoparib 1 mg/day for 24 cycles (28 days per cycle), continuing until withdrawn or discontinued, eg, until RECIST 1.1 progression or unacceptable toxicity.
  Interventions: Drug: Talazoparib Tosylate

INTERVENTIONS:
Drug: Talazoparib Tosylate — Talazoparib1 mg/day is to be administered orally on a continuous dosing schedule.
  Other Names: Talzenna; BMN-673

SUMMARY:
This purpose of this study is to test if talazoparib is safe and evaluate its response to advanced breast cancer associated with mutation of gene called PALB.

DETAILED DESCRIPTION:
Primary Objectives: To evaluate whether talazoparib monotherapy can induce a 30% rate of objective response in subjects with advanced breast cancer associated with a PALB2 mutation.

Secondary Objective(s)

1. To evaluate the safety of talazoparib in subjects with advanced PALB2 mutation associated breast cancer
2. To evaluate the progression free survival (PFS) of talazoparib monotherapy in subjects with advanced PALB2 mutation associated breast cancer
3. To evaluate the clinical benefit rate (CBR) of talazoparib monotherapy in subjects with advanced PALB2 mutation associated breast cancer
4. To evaluate the ability of circulating tumor DNA (ctDNA) to identify and characterize the nature of PALB2 mutations at baseline and upon progression in subjects with advanced PALB2 mutation associated breast cancer treated with talazoparib monotherapy
5. To evaluate patient reported quality of life on talazoparib monotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic or recurrent HER2 negative breast cancer (IHC or fluorescence in situ hybridization (FISH) per ASCO/CAP guidelines).
2. Deleterious or suspected deleterious mutation in PALB2 assessed by Clinical Laboratory Improvement Amendments (CLIA) approved tumor next generation sequencing (NGS) or germline assay.
3. Women and men ≥ 18 years of age.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
5. All clinically significant toxic effects of prior cancer therapy resolved to Grade ≤ 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE, v 5.0), except alopecia and G2 neuropathy.
6. Measurable disease per RECIST v1.115 (CT CAP with contrast and bone scan or positron emission tomography computer tomography (PET/CT) with IV contrast needed within 28 days of Cycle 1 Day 1. If patients have a history of brain metastases, a MRI brain or CT head with contrast is required).
7. A minimum 21 day wash out from previous treatment is required.
8. No evidence of progression on platinum (e.g., carboplatin or cisplatin) or within 8 weeks of last platinum dose
9. Adequate hematologic function

   * Absolute neutrophil count (ANC) ≥ 1,500 cells/μL (≥ 1,500/mm3)
   * Hemoglobin ≥ 9.0 g/dL with last transfusion at least 14 days before Day 1 of study drug
   * Platelets ≥ 100,000 cells/μL (≥ 100,000/mm3)
10. Adequate hepatic function

    * Bilirubin ≤ 1.5 times the specific institutional upper limit of normal (ULN). Exception: If Gilbert's syndrome; then ≤ 5 times ULN.
    * Aspartate transaminase (AST) and alanine transaminase (ALT) each ≤ 2.5 x ULN; if liver function abnormalities are due to hepatic metastasis, then AST and ALT ≤ 5 x ULN
11. Adequate renal function

    * Serum creatinine ≤ 1.5 x ULN; or
    * Calculated creatinine clearance > 50 mL/min using the Cockcroft Gault formula.
12. Able to take oral medications
13. Received 0 3 prior therapies for advanced disease
14. Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test and be willing to have additional urine pregnancy tests during the study. Women considered not of childbearing potential include those who have had no menstrual period for at least 1 year and have an estradiol in the postmenopausal range, or had tubal ligation at least 1 year prior to screening, or who have had total hysterectomy or bilateral oophorectomy.
15. WOCBP must agree to use effective contraception as of C1D1 and for 3 months after the last dose.
16. Male participants and their female partners of child bearing potential must be willing to use an appropriate method of contraception during the study and for 3 months after the last dose.
17. Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research related procedures
18. Willing and able to comply with all study procedures
19. Adequate archival or fresh tumor sample from metastatic biopsy site; archival tumor from the primary breast tumor may be submitted if metastatic biopsy is not available and/or infeasible

Exclusion Criteria:

1. Breast cancer amenable to curative treatment.
2. Prior treatment with a PARP inhibitor.
3. Deleterious or suspected deleterious germline or somatic BRCA1 or BRCA2 gene mutation. Patients with variants of unknown significance will be eligible.
4. Active Brain metastases OR leptomeningeal carcinomatosis. EXCEPTION: Adequately treated brain metastases documented by baseline CT or MRI scan that have not progressed since previous scans and do not require corticosteroids (prednisone 5 mg/day or equivalent allowed) for management of central nervous system (CNS) symptoms. A repeat CT or MRI following the identification of CNS metastases (obtained at least 2 weeks after definitive therapy) must document adequately treated brain metastases.
5. Pregnant or breastfeeding patients.
6. Other malignancy that is either active or for which patient has received treatment in the last three years excluding non melanoma skin cancer and carcinoma in situ of the cervix or breast.
7. Known active hepatitis B or hepatitis C.
8. Investigational agents within 28 days of C1D1.
9. Radiation therapy within 14 days of C1D1.
10. Major surgery within 21 days of C1D1.
11. Concurrent disease or condition that would interfere with study participation or safety, such as any of the following:

    a. Active, clinically significant infection either grade > 2 by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 or requiring the use of parenteral anti microbial agents within 7 days of C1D1.
12. Clinically significant bleeding diathesis or coagulopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 8 weeks +/-1 week
  Response to treatment will be assessed as the number and proportion of participants who achieve either a confirmed complete response (CR) or partial response (PR). The outcome is reported as numbers without dispersion. Clinical response will be assessed as follows.
  CR: Complete disappearance of all clinical evidence of disease PR: Decrease in size or amount of measurable disease lesions Progressive disease (PD): Worsening of lesions; appearance of new lesions; or recurrence of lesions Stable disease (SD): Disease status that is neither CR, PR, nor PD.

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) | 8 weeks +/- 1 week
  Clinical benefit rate (CBR) will be reported as the number and proportion of participants who achieve CR, PR or Stable Disease (SD) 6 months. The outcome is reported as numbers without dispersion.
Progression-free survival (PFS) | 8 weeks +/- 1 week
  Median progression free survival (PFS) will be assessed as the period of survival from therapy initiation without the development of progressive disease per RECIST 1.1. The outcome is reported as a number without dispersion.
Patient-reported Quality of Life (QoL) | 8 weeks +/- 1 week
  Change from Baseline in Global Health Status/Quality of Life (QoL) Measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ C30) EORTC QLQ C30 has 30 questions. First 28 questions evaluate 5 functional scales and 3 symptom scales and other single items. Each question assessed on 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much); functional scales: higher score = better level of functioning; symptom scale: higher score = more severe symptoms; for single items: higher score= more severe problem. Last 2 questions evaluate global health status (GHS)/QoL. Each question is assessed on 7 point scale (1=very poor to 7=excellent). Scores averaged, transformed to 0-100 scale; higher score means a better quality of life/better level of functioning. The outcome will be reported as the median QoL score with standard deviation.
Number of participants with Treatment-related Adverse Events ≥ Grade 3 | 3 years
  Toxicity will be assessed as adverse events that are severe or greater (≥ Grade 3), and possibly, probably, or definitely related to talazoparib. The outcome will be reported as the total number of qualifying events, a number without dispersion.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Telli, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No